CLINICAL TRIAL: NCT06406790
Title: A Multicenter, Single-Blind, Prospective Randomized Post-Approval Study Comparing the Safety and Effectiveness of CraniSeal Dural Sealant to DuraSeal Dural Sealant for Dural Sealing in Elective Cranial Surgery
Brief Title: CraniSeal Post Approval Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pramand LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRA-CT-0003
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Leak, Cerebrospinal Fluid
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 CraniSeal vs Comparator
Who Masked: Participant
Masking Description: Participant will be blinded to dural sealant until they have completed 90 day study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CraniSeal (Experimental): CraniSeal
  Interventions: Device: CraniSeal
- DuraSeal (Active Comparator): DuraSeal
  Interventions: Device: DuraSeal

INTERVENTIONS:
Device: CraniSeal — CraniSeal is a PEG Dural Sealant
  Arms: CraniSeal
Device: DuraSeal — DuraSeal is a PEG Dural Sealant
  Arms: DuraSeal

SUMMARY:
To collect post-approval data comparing the safety and effectiveness of CraniSeal Dural Sealant to DuraSeal Dural Sealant. The study has been powered specifically to determine whether the CraniSeal device when used as an adjunct to sutured dural closure following elective cranial surgery is no worse than (i.e., non-inferior) to the DuraSeal device with respect to proportion of subjects free from post-operative cerebrospinal fluid (CSF) leaks. Additional safety outcomes (i.e., surgical site infections and adverse events/device-related adverse events) will also be captured and compared.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Patient is scheduled for an elective infratentorial or supratentorial cranial procedure under general anesthesia that entails a dural incision
3. Patient requires a procedure involving surgical wound classification Class I/Clean
4. Patient signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedures.
5. Patients who are able to comply with study requirements.

General Exclusion Criteria:

1. Patient requires a procedure involving translabyrinthine, transsphenoidal, transoral and/ or any procedure that penetrates the air sinus or mastoid air cells; superficial penetration of air cells are not excluded
2. Patient has had a prior intracranial neurosurgical procedure in the same anatomical location
3. Patient with diagnosis of severely altered renal (creatinine levels > 2.0 mg/dL) or hepatic (total bilirubin > 2.5 mg/dL) function
4. Patient diagnosed with a compromised immune system or autoimmune disease (WBC count less than 4000/uL or greater than 20,000/uL)
5. Patients undergoing cranial procedures involving petrous bone drilling
6. Patients with traumatic injuries to the head or dural disease in planned dural closure area
7. Patients who are pregnant or lactating
8. Patient with an active infection
9. Patient is undergoing cranial procedures involving non-autologous duraplasty material that are not collagen based
10. Patients requiring re-opening of planned surgical area within 90 days after surgery.
11. Patient with a known allergy to FD&C Blue #1 dye
12. Patient is not able to tolerate multiple Valsalva maneuvers, or transient elevation of CSF pressure during Valsalva maneuvers is not possible (e.g. the presence of a temporary or permanent CSF shunt
13. Presence of hydrocephalus
14. Patient with a diagnosis of uncontrolled diabetes (e.g., persistent HbA1c elevation of >9% despite standard diabetes care),
15. Patient has a documented, uncorrectable clinically significant coagulopathy (e.g., PTT>37 seconds or INR >1.5 units)
16. Patient is not likely to comply with the follow-up evaluation schedule.
17. Contraindications to both an MRI and CT scan.
18. Patients participating in any investigational device study within 30 days or currently receiving an investigational drug/biologic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Absence of CSF Leaks | 90 days
  absence of CSF leaks on study

OTHER OUTCOMES:
TEAEs and TESAEs | 90 days
  treatment emergent events on study

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Keck Medical Center at USC, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Jacobs Institute, Buffalo, New York
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No